CLINICAL TRIAL: NCT01835067
Title: Intravitreal Tissue Plasminogen Activator And Perfluoropropane for Neovascular Age-related Macular Degeneration With Associated Submacular Haemorrhage: a Multi-centre, Randomized, Double-masked, Sham-controlled, Factorial, Feasibility Study
Brief Title: Intravitreal tPA and C3F8 for the Treatment of Submacular Haemorrhage as a Complication of Neovascular AMD
Acronym: TAPAS
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: King's College Hospital NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: EudraCT Number: 2012-004078-24
Record Dates: First submitted 2013-04-16; First posted 2013-04-18 (Estimated); Last update posted 2020-07-14 (Actual); Status verified 2020-02

CONDITIONS: Exudative Macular Degeneration; Retinal Hemorrhage
Keywords: Macular degeneration; Submacular haemorrhage
MeSH Terms: conditions — Wet Macular Degeneration; Retinal Hemorrhage; Macular Degeneration | interventions — Ranibizumab; perflutren; Tissue Plasminogen Activator

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Control Group (A) (Sham Comparator): Ranibizumab only (active control). Participants will receive a 'sham injection' to simulate C3F8 and/or tPA administration.
  Interventions: Drug: Ranibizumab
- C3F8 Only Group (B) (Experimental): C3F8 given. Ranibizumab given as standard.
  Interventions: Drug: Ranibizumab; Drug: C3F8 Gas
- tPA and C3F8 Group (C) (Experimental): Both C3F8 gas and tPA given. Ranibizumab given as standard.
  Interventions: Drug: Ranibizumab; Drug: C3F8 Gas; Drug: tPA
- tPA Only Group (D) (Experimental): tPA given. Ranibizumab given as standard.
  Interventions: Drug: Ranibizumab; Drug: tPA

INTERVENTIONS:
Drug: Ranibizumab — Single intravitreal injection of 500 micrograms ranibizumab in 0.05mls
  Other Names: Lucentis®
Drug: C3F8 Gas — Single intravitreal injection of 0.3 mls C3F8
  Other Names: Perfluoropropane; Perflutren; Octafluoropropane
  Arms: C3F8 Only Group (B); tPA and C3F8 Group (C)
Drug: tPA — Single intravitreal injection of 50 micrograms tPA in 0.05 mls
  Other Names: tissue plasminogen activator; alteplase; Actilyse®
  Arms: tPA Only Group (D); tPA and C3F8 Group (C)

SUMMARY:
This study will recruit patients who have recently had a submacular haemorrhage (bleed under the part of the retina responsible for detailed vision), as a complication of wet age-related macular degeneration (wet AMD). Wet AMD is a very common disease where abnormal blood vessels form under the retina and leak, causing a significant reduction in vision.

The study will investigate treatment of the bleed with various combinations of the two drugs: tissue plasminogen activator (tPA) - designed to dissolve the blood clot; and perfluoropropane (C3F8) - designed to shift the blood clot away from the central part of the retina (the macula). tPA is a commonly used 'clot-buster' drug for the treatment of stroke. C3F8 is a gas commonly used in eye surgery. Patients recruited will be divided into four groups: control group that receive none of the above drugs; one group that receives only tPA; one group that receives only C3F8; and one group that receives both.

All patients will receive the current gold standard treatment for wet AMD, ranibizumab (Lucentis®).

The aim of the study is to improve vision in a condition, which left untreated, would cause severe visual loss.

DETAILED DESCRIPTION:
Age-related macular degeneration (AMD) is the commonest cause of blindness worldwide. Its prevalence increases with age, being relatively rare under 60 years and reaching its peak incidence in those older than 80 years. AMD principally affects central vision, which is responsible for the ability to see fine detail and the disease rapidly destroys the ability to read normal print, recognise faces, drive, and watch television. It can therefore have a profound effect on quality of life.

There are two main forms of AMD; the dry form, in which there is slow degeneration of the cells responsible for sight, resulting in gradual visual loss; and the wet form (neovascular), which occurs when abnormal blood vessels (choroidal neovascularisation) grow under the retina, the part of the eye which is responsible for sensing light, like the film of a camera. These new blood vessels have weak walls leading to leakage of fluid (oedema), and sometimes significant amounts of bleeding (submacular haemorrhage - SMH). These rapidly lead to central visual distortion and blurring. Although the dry form is commoner, the wet form more commonly results in profound central visual loss and is responsible for the majority of cases that ultimately require blind registration.

The current best treatment ('gold-standard') for wet AMD is the drug ranibizumab (Lucentis®), which aims to shrink and destroy the abnormal blood vessels responsible for the visual symptoms. In several trials ranibizumab has been shown to improve vision in patients with wet AMD.

It is not uncommon for patients with wet AMD to develop SMH, which when it occurs, significantly reduces the patient's visual prognosis. SMH is thought to have a number of toxic consequences on the retinal function.

This study investigates the use of two drugs: tissue plasminogen activator (tPA), a 'clot-buster' drug used to treat stroke, which is designed to dissolve the clot over the central retina (macula); and perfluoropropane (C3F8), a gas commonly used in retinal surgery, which is designed to displace the clot away from the macula.

This study is a randomized, double-masked, clinical trial with a recruitment target of 55 people with SMH and wet AMD. Participants will be allocated to one of four groups; a control group receiving none of the above drugs; one group receiving only tPA; one group receiving only C3F8; and one group receiving both. All patients will receive the 'gold-standard' treatment of ranibizumab for their underlying wet AMD. We aim to determine if tPA and/or C3F8 produce a visual outcome that is superior to standard care, with a favourable safety profile. We will also measure the size of the blood clot and scarring using computer analysis of macula photographs.

ELIGIBILITY:
Inclusion criteria:

* Adults of either sex aged 50 years and older;
* SMH associated with treatment-naive or previously treated wet AMD, including retinal angiomatous proliferation (RAP) and idiopathic polypoidal choroidal vasculopathy (IPCV);
* SMH of at least 1 disc area, involving the fovea, and of sufficient density to obscure RPE detail;
* Written informed consent to participate in the study.Only one eye will be eligible for inclusion in this study.

Exclusion criteria:

* SMH that is known to have been present for greater than 2 weeks duration, as evidenced by history, pre-trial documentation, or fundus appearance;
* Presence of significant vitreous haemorrhage precluding accurate retinal assessment in the study eye;
* Diabetic maculopathy in the study eye;
* Visually significant cataract in the study eye;
* Amblyopia in the study eye;
* Presence of other ocular disease causing concurrent vision loss in the study eye;
* Advanced glaucoma in the study eye (cup-to-disc ratio greater than 0.8);
* Pregnant and or lactating women;
* Women of childbearing potential including those who are not sterilised or at least one year post menopausal;
* Participation in a clinical interventional trial in the preceding 6 months;
* Documented evidence of a visual acuity less than 25 ETDRS letters at three consecutive visits in the study eye, prior to the onset of submacular haemorrhage;
* Participants who are known to have been ineligible for NICE approved ranibizumab therapy prior to the development of the SMH;
* Current treatment for wet age-related macular degeneration with an intravitreal agent other than ranibizumab, bevacizumab or aflibercept;
* Patients who, in the opinion of the Investigator, would not be willing or able to comply with the study protocol, including posturing requirements.
* Patients who show insufficient understanding of the clinical trial or treatment options.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2019-11 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Mean ETDRS visual acuity | 3 months

SECONDARY OUTCOMES:
Mean ETDRS visual acuity | 1 and 12 months
Percentage patients 15 letters or greater improvement in ETDRS visual acuity | 12 months
Percentage patients 0 letters or greater improvement in ETDRS visual acuity | 12 months
Percentage patients 15 letters or greater loss in ETDRS visual acuity | 12 months
Mean total area of macular haemorrhage on colour fundus photography | 1, 3 and 6 months
Greatest linear dimension of macular haemorrhage on colour fundus photography | 1, 3 and 6 months
Presence of subfoveal blood on colour fundus photography | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Timothy L Jackson, PhD,FRCOpht, Principal Investigator — King's College Hospital NHS Trust
Locations (5):
- United Kingdom (5):
  - Maidstone Hospital, Maidstone, Kent
  - Sunderland Eye Infimary, Sunderland, Tyne and Wear
  - Hull & East Yorkshire Hospital NHS Trust, Hull
  - King's College Hospital NHS Foundation Trust, London
  - Southend University Hospital NHS Foundation Trust, Southend

IPD SHARING:
Plan to Share IPD: Undecided
The Investigator(s) and the institution(s) shall permit trial-related monitoring, audits, REC review, and regulatory inspections (where appropriate) by providing the Sponsors, Regulators and REC direct access to source data and other documents (i.e. patients' case sheets, blood test reports, X-ray reports, histology reports etc). Where necessary, inspection may also take place at the site's facilities.

REFERENCES:
- [Derived] Murphy GSP, Saleh A, Ayis S, Cheema MR, Mehta A, Steel DH, Membrey L, Costen M, Jackson TL. Tissue Plasminogen Activator or Perfluoropropane for Submacular Hemorrhage in Age-Related Macular Degeneration: A Factorial Randomized Clinical Trial. JAMA Ophthalmol. 2024 Dec 1;142(12):1157-1164. doi: 10.1001/jamaophthalmol.2024.4297. PMID 39418015